CLINICAL TRIAL: NCT06677931
Title: Safety and Efficacy of Umbilical Cord Mesenchymal Stem Cell-Derived Exosomes in the Treatment of Melasma, a Prospective, Randomized, Controlled Clinical Trial
Brief Title: Umbilical Cord Mesenchymal Stem Cell-Derived Exosomes in the Treatment of Melasma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Principal Investigator, ChenXiaosong, professor, Fujian Medical University Union Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024YF028-01
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-06

CONDITIONS: Melasma
Keywords: Melasma; stem cell; exosomes
MeSH Terms: conditions — Melanosis | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1565 non-ablative fractional laser combined with normal Saline (Placebo Comparator): 1565 non-ablative fractional laser combined with normal Saline
  Interventions: Procedure: Placebo Comparator:1565 non-ablative fractional laser combined with normal Saline
- 1565 non-ablative fractional laser combined with umbilical cord mesenchymal stem cell exosomes (Experimental): 1565 non-ablative fractional laser combined with umbilical cord mesenchymal stem cell exosomes
  Interventions: Procedure: 1565 non-ablative fractional laser combined with umbilical cord mesenchymal stem cell-derived exosomes.

INTERVENTIONS:
Procedure: Placebo Comparator:1565 non-ablative fractional laser combined with normal Saline — Based on the patient's age, skin color, location of skin lesions, and Fitzpatrick skin type, adjust treatment parameters accordingly. The operator holds the treatment head, vertically applies parallel sweeps closely to the lesion area until the endpoint of slight skin redness is reached. After completion, apply normal Saline.
  Arms: 1565 non-ablative fractional laser combined with normal Saline
Procedure: 1565 non-ablative fractional laser combined with umbilical cord mesenchymal stem cell-derived exosomes. — Based on the patient's age, skin color, location of skin lesions, and Fitzpatrick skin type, adjust treatment parameters accordingly. The operator holds the treatment head, vertically applies parallel sweeps closely to the lesion area until the endpoint of slight skin redness is reached. After completion, apply exosomes.
  Arms: 1565 non-ablative fractional laser combined with umbilical cord mesenchymal stem cell exosomes

SUMMARY:
Melasma is a refractory skin disease with a complex pathogenesis and difficult treatment. Research has found that mesenchymal stem cell-derived exosomes have effects such as anti-wrinkle formation, anti-inflammation, antioxidant properties, skin whitening, and promotion of skin regeneration. Recent studies show that there is damage to the basement membrane in melasma skin lesions, and the regenerative repair function of mesenchymal stem cell-derived exosomes can repair the damaged basement membrane in melasma skin lesions, thereby effectively treating melasma. This study aims to observe the therapeutic effect of umbilical cord mesenchymal stem cell-derived exosomes combined with 1565 non-ablative fractional laser treatment for melasma, verify the enhancement effect of 1565 non-ablative fractional laser, and also explore a new combined treatment method for melasma that is effective, low in side effects, low in recurrence rate, and provides good patient comfort.

DETAILED DESCRIPTION:
Exosomes are small, uniform lipid bilayer vesicles with a molecular diameter of 30-150 nanometers, formed by cells and actively secreted into the extracellular space. They contain proteins, peptides, lipids, nucleic acids, growth factors, hormones, and other substances. Exosomes derived from stem cells share similar functions with stem cells, including tissue repair and regeneration, enhancing the survival of transplanted fat, anti-inflammatory, and antioxidant effects. Compared to stem cells, exosomes are more stable, easier to preserve, manage, and control, and their content can be manipulated in terms of type and quantity. They lack live cells and have low immunogenicity. Research has found that stem cell-derived exosomes have various effects in anti-aging and medical aesthetics.

Melasma is an acquired pigmentation disorder predominantly affecting females. Its pathogenesis is complex, and treatment is challenging, making it one of the refractory skin diseases. Current treatment methods have long treatment cycles, high recurrence rates, and poor patient compliance, with treatment outcomes still not ideal. Recent studies show damage to the basement membrane in melasma skin lesions, and the regenerative repair function of stem cell-derived exosomes can repair the damaged basement membrane in these lesions, thus effectively treating melasma.

Due to the skin's barrier function, exosomes from stem cells can hardly penetrate the skin barrier. In recent years, various physicochemical methods such as chemical enhancers, nanotechnology, ultrasound, microneedles, radiofrequency, or thermal ablation have been introduced to facilitate the transdermal delivery of biologics. However, they pose significant issues in terms of skin irritation and damage while aiding in overcoming the skin barrier for effective enhancement. Therefore, finding methods that are minimally irritating to the skin and capable of facilitating the transdermal delivery of biologics remains a challenge in transdermal drug delivery.

This study aims to observe the therapeutic effect of umbilical cord mesenchymal stem cell-derived exosomes combined with 1565 non-ablative fractional laser treatment for melasma, validate the enhancement effect of 1565 non-ablative fractional laser, and explore a new combined treatment method for melasma that is effective, low in side effects, low in recurrence rate, and provides good patient comfort.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 60 years with good overall health.
2. Diagnosed with melasma according to clinical diagnostic criteria and efficacy standards (revised edition), with facial skin lesions.
3. Fully understands and comprehends the content and significance of the study, implementation plan, potential benefits, risks, mitigation measures, participant rights and obligations (including privacy protection and voluntary withdrawal), and willingly signs the informed consent form to participate in the clinical study, and can cooperate well.
4. Exclusion of inflammatory post-pigmentary disorders, malar melasma, Riehl's melanosis, pigmentary lichenoid dermatosis, and other skin diseases.
5. Agrees not to use other cosmetic treatments related to the study during the research period.

Exclusion Criteria:

1. Patients who refuse to sign the informed consent form to participate in the trial.
2. History of significant organ diseases, autoimmune diseases, or immune dysfunction.
3. Abnormal coagulation function, current use of anticoagulants, tendency for thrombosis, or family history of genetic diseases.
4. Pregnant or lactating women.
5. Patients who have taken oral contraceptives or hormone replacement therapy during the study period or in the past 12 months.
6. Patients with a keloid-prone constitution.
7. Locally damaged or actively affected by other skin diseases.
8. History of severe multiple allergies, genetic allergies, photosensitivity or history of photosensitive drugs such as sulfonamides and tetracyclines, allergy to local anesthetics, lidocaine components, or planned desensitization therapy during the study.
9. History of post-inflammatory hyperpigmentation.
10. Previously treated for melasma.
11. Previous chemical peels, abrasion procedures, or other resurfacing treatments on the face.
12. Chronic skin diseases, especially infectious, allergic, and inflammatory systemic skin diseases such as widespread eczema, pemphigus, pemphigoid, etc.
13. Patients currently participating in other clinical studies.
14. Other reasons deemed unsuitable for the clinical study by the investigator.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-08-28 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
melasma area and severity index, MASI | 1, 2, 3, 4, 5, 6, 7, 8 months after the first treatment
  MASI = 0.3(DMR + HMR)AMR + 0.3(DF + HF)AF + 0.3(DML + HML)AML + 0.1(DC + HC)AC, The total score is 48 points, with lower scores indicating less severity of melasma. MASI is jointly assessed by two physicians from this department, taking the average value. If there is a significant difference in the evaluation results of the two physicians, a third physician from the same department will be consulted, and the average value of the two closest assessments will be taken.

SECONDARY OUTCOMES:
physician's global assessment, PGA | 1, 2, 3, 4, 5, 6, 7, 8 months after the first treatment
  Based on the residual condition of pigmented lesions after treatment, a score of 0 to 6 is assigned: 0 points for complete clearance (100%) or only minimal residual pigmentation, 1 point for essentially cleared (≥ 90%), 2 points for marked improvement (75% ~ 89%), 3 points for moderate improvement (50% ~ 74%), 4 points for slight improvement (25% ~ 49%), 5 points for no improvement (< 25%), 6 points for worsening compared to before treatment.
Patient satisfaction evaluation | 1, 2, 3, 4, 5, 6, 7, 8 months after the first treatment
  Patient satisfaction is evaluated using a self-assessment satisfaction scale. It is divided into very satisfied (improvement ≥ 75%), satisfied (improvement 50% ~ 75%), average (improvement 25% ~ 49%), and dissatisfied (improvement ≤ 25%); Satisfaction rate = (Number of very satisfied cases + Number of satisfied cases) / Total number of cases × 100%.
Occurrence of adverse reactions | 1, 2, 3, 4, 5, 6, 7, 8 months after the first treatment
  Observation of adverse reactions including erythema, burning, itching, dryness, irritation, hyperpigmentation, edema, scar formation, skin breakdown, and skin infection.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Affiliated Union Hospital of Fujian Medical University, Fuzhou, Fujian
  - Chenxiaosong, Fujian, Fuzhou